CLINICAL TRIAL: NCT05935371
Title: The Impact of Severe Perineal Trauma on Maternal Mental Health and Intra-family Relationships
Brief Title: Consequences of Obstetric Anal Sphincter Injuries on Maternal Psychology and Relationship Experience
Acronym: COMPaRE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: London North West Healthcare NHS Trust (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 327802
Record Dates: First submitted 2023-06-04; First posted 2023-07-07 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-06

CONDITIONS: Obstetric Complication; Obstetric Trauma; Perineal Tear; Incontinence; Mental Health Impairment; Relation, Family; Relation, Mother-Child

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group - women with obstetric anal sphincter injuries: * Adult women who have had a vaginal delivery
  * ≥ 18 years
  * Capacity to consent
  * English-speaking
  * Primiparous/multi-parous
- Control group - women without perineal tears: * Adult women who have had a vaginal delivery
  * ≥ 18 years
  * Capacity to consent
  * English-speaking
  * Primiparous/multi-parous

SUMMARY:
The aim is to ascertain whether sustaining an Obstetric Anal Sphincter Injury negatively impacts intra-family relationships and increases the risk of mental health conditions, including a women's perception of herself and her self-esteem. Research in this field will ensure that the correct care and adequate support is provided for these patients in the post-natal period and beyond. Recognition of these conditions and the provision of support for these patients may improve relationships, leading to improved parenting and positive outcomes for the child. It ought to be highlighted that the sequelae of obstetric anal sphincter injuries, including anal incontinence, may manifest later on in the female life course and therefore life-long accessibility to help and therapies is advocated for these women.

DETAILED DESCRIPTION:
Obstetric anal sphincter injuries encompass grade 3 and 4 perineal tears and effect the integrity of the anorectal sphincter complex, with or without involvement of the anorectal mucosa. Obstetric anal sphincter injuries occur following a vaginal delivery and are more common in primiparae women, occurring with an incidence in the UK of 6.1% compared to 1.7% in those who are multiparae. Although obstetric anal sphincter injuries is fairly uncommon, the rate of these injuries in singleton, cephalic and first vaginal deliveries, has reportedly tripled from 1.8% to 5.9% from 2000 to 2012. This may, however, be secondary to better detection of these injuries following improvements in education, training and the utilization of a standardized classification system for perineal tears. To address the rising obstetric anal sphincter injury rates, the obstetric anal sphincter injury care bundle was introduced which primarily focused on interventions in the antenatal period to reduce the incidence of these injuries. Prevention of these injuries, however, will not always be possible, even with the best efforts of care. Therefore, focus should also be placed on the optimal management of these patients post-partum. This is especially important as these injuries may be associated with a myriad of devastating and stigmatizing sequelae, including faecal and urinary incontinence, dyspareunia, rectovaginal fistulae, perineal pain and pelvic organ prolapse. It is not surprising, therefore, that sustaining such an injury may impact a woman's decision to have another baby. Severe perineal trauma, with or without complications may, understandably, cause a negative impact on the mental health of afflicted mothers.

Suffering from the complications of these injuries may impact on an individual's quality of life and day-to-day functioning, further augmenting the psychological impact of obstetric anal sphincter injuries. Research has highlighted obstetric anal sphincter injuries to be a risk factor for the development of post traumatic stress disorder symptoms. At present, mothers with these injuries are not routinely screened for these conditions in the post-natal period. Preliminary research has shown that acquiring such an injury negatively affects the relationship between a mother and her child, which invariably has a deleterious effect on a child's development.

This study delivers a questionnaire which incorporates existing, screening tools including the Patient Health Questionnaire-9 (PHQ-9), Generalised Anxiety Disorder-7 (GAD-7), Post-traumatic stress disorder checklist (PCL-5), Rosenberg self-esteem score, Arizona sexual experiences scale, Dyadic Adjustment Scale and the Mother infant bonding scale (MIBS) to assess the impact of these injuries on a women's mental health and intra-family relationships. The PHQ-9 has been shown to be on par with the Edinburgh postnatal depression scale in screening for depression in the perinatal period.

Recognition of mental health dysfunction within this cohort, if present, would facilitate early intervention which may in turn reduce the long-term consequences of a traumatic child birth.

ELIGIBILITY:
Inclusion Criteria:

* as aforementioned previously

  * Adult women who have had a vaginal delivery
  * ≥ 18 years
  * Capacity to consent
  * English-speaking
  * Primiparous/multi-parous

Exclusion Criteria:

* Women who have had a caesarean section
* Women who are unable to consent
* Patient who do not speak English

Ages: 18 Years to 60 Years | Sex: Female
Age Groups: Adult
Study Population: English-speaking women, over the age of 18, with capacity to consent (able to comprehend and retain information, weight out the risks and benefits and communicate a decision back to the researcher) and who have had a vaginal delivery are eligible to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Estimated)
Dates: Start 2023-10-26 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
the impact of an obstetric anal sphincter injury on | study to be completed within 12 months
  the incidence of depression using the patient health questionnaire-9 screening tool. The binary outcome cut off is 10 for this questionnaire. The higher the score the worse the outcome. Mininum score 0. Maximum score 27.
the impact of an obstetric anal sphincter injury on | study to be completed within 12 months
  the presence and severity of post-traumatic stress disorder using the post-traumatic stress disorder checklist (PCL-5) screening tool. Outcome is continuous. The higher the score, the worse the outcome. Minimum score 0. Maximum score 80.
the impact of an obstetric anal sphincter injury on | study to be completed within 12 months
  patient self-esteem using the rosenberg self-esteem scale. The binary outcome cut off is 15. Range is 0-30. Scores below 15 suggest low self esteem.
the impact of an obstetric anal sphincter injury on | study to be completed within 12 months
  sexual dysfunction (quantifying sex drive, arousal, vaginal lubrication/penile erection, ability to reach and satisfaction from orgasm) using the arizona sexual experiences scale. Range of score from 5-30. A total score > or equal to 19 or any 1 item with an individual score of more than or equal to 5 or any 3 items with individual scores of more than or equal to 4 are highly correlated with the presence of sexual dysfunction.
the impact of an obstetric anal sphincter injury on | study to be completed within 12 months
  quality of a relationship within an intact couple using the abbreviated dyadic adjustment scale (DAS-4). A score of 14 is the binary outcome cut off.0-21 range. Higher the score the better the relationship.
the impact of an obstetric anal sphincter injury on | study to be completed within 12 months
  anxiety using the generalised anxiety disorder-7 screening tool. The binary outcome cut off is 10. Range is 0-21. The higher the score, the greater the anxiety.
the impact of an obstetric anal sphincter injury on | study to be completed within 12 months
  mother to infant bonding using the mother to infant bonding scale. Range score 0-24. The higher the score, the more likely bonding is disrupted.

SECONDARY OUTCOMES:
The influence of the following factor in predicting severity and risk of mental health disorders and relationship dysfunction (specifically pertaining to relationship with partner and child): | study to be completed over a 12 month period
  age
The influence of the following factor in predicting severity and risk of mental health disorders and relationship dysfunction (specifically pertaining to relationship with partner and child): | study to be completed over a 12 month period
  type of delivery (e.g. instrumental/assisted or spontaneous vaginal delivery)
The influence of the following factor in predicting severity and risk of mental health disorders and relationship dysfunction (specifically pertaining to relationship with partner and child): | study to be completed over a 12 month period
  number of vaginal births
The influence of the following factor in predicting severity and risk of mental health disorders and relationship dysfunction (specifically pertaining to relationship with partner and child): | study to be completed over a 12 month period
  history of previous obstetric anal sphincter injury. The researchers will attempt to obtain this information by reviewing the patient's medical records and asking the patient if they have been previously diagnosed with an obstetric anal sphincter injury.
The influence of the following factor in predicting severity and risk of mental health disorders and relationship dysfunction (specifically pertaining to relationship with partner and child): | study to be completed over a 12 month period
  grade of tear (assessed clinically or radiologically)
The influence of the following factor in predicting severity and risk of mental health disorders and relationship dysfunction (specifically pertaining to relationship with partner and child): | study to be completed over a 12 month period
  Obstetric Anal sphincter Injury (OASI) induced incontinence and severity (as assessed by St Mark's incontinence scale). St Mark's score ranges from 0-24. Abnormal is scores more than 5. The greater the score, the greater the incontinence score.

CONTACTS AND LOCATIONS:
Locations (1):
- London Northwest Healthcare NHS Trust, London, Brent, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Skari H, Skreden M, Malt UF, Dalholt M, Ostensen AB, Egeland T, Emblem R. Comparative levels of psychological distress, stress symptoms, depression and anxiety after childbirth--a prospective population-based study of mothers and fathers. BJOG. 2002 Oct;109(10):1154-63. doi: 10.1111/j.1471-0528.2002.00468.x. PMID 12387470
- [Background] Ertan D, Hingray C, Burlacu E, Sterle A, El-Hage W. Post-traumatic stress disorder following childbirth. BMC Psychiatry. 2021 Mar 16;21(1):155. doi: 10.1186/s12888-021-03158-6. PMID 33726703
- [Background] Thornton C, Schmied V, Dennis CL, Barnett B, Dahlen HG. Maternal deaths in NSW (2000-2006) from nonmedical causes (suicide and trauma) in the first year following birth. Biomed Res Int. 2013;2013:623743. doi: 10.1155/2013/623743. Epub 2013 Aug 19. PMID 24024205
- [Background] Garthus-Niegel S, Horsch A, Handtke E, von Soest T, Ayers S, Weidner K, Eberhard-Gran M. The Impact of Postpartum Posttraumatic Stress and Depression Symptoms on Couples' Relationship Satisfaction: A Population-Based Prospective Study. Front Psychol. 2018 Sep 19;9:1728. doi: 10.3389/fpsyg.2018.01728. eCollection 2018. PMID 30283380
- [Background] Bick Obe D, Hall J, Keighley MRB. The impact of severe perineal trauma on a woman's relationship with her child: a hidden consequence. Midwifery. 2022 May;108:103323. doi: 10.1016/j.midw.2022.103323. Epub 2022 Mar 22. No abstract available. PMID 35366595
- [Background] Shonkoff M, Duncan GJ, Yoshikawa H, et al. Maternal depression can undermine the development of young children. Centre on the developing child, Harvard University; 2009.
- [Background] Sabourin S, Valois P, Lussier Y. Development and validation of a brief version of the dyadic adjustment scale with a nonparametric item analysis model. Psychol Assess. 2005 Mar;17(1):15-27. doi: 10.1037/1040-3590.17.1.15. PMID 15769225